CLINICAL TRIAL: NCT03981471
Title: STrategies and mechAnisms of Community-Based falL Prevention in Elderly
Brief Title: Fall Prevention in Elderly: Mechanisms and Strategies
Acronym: STABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Rehabilitation Technical Aids (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Pengxu Wei, Director, National Research Center for Rehabilitation Technical Aids
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018YFC2001401
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Elderly
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly without fall history (Other): Elderly people in the community who have no fall history
  Interventions: Behavioral: Exercise
- Elderly with fall history (Other): Elderly people in the community who have fall history
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Elderly people with or without fall history receive exercise to improve balance. Exercise interevention will be given 6 months in 2020. Outcomes (incidence of fall and biological tests) between two arms will be compared.

SUMMARY:
In communities with over 100,000 residents, to investigate the incidence and mechanisms of fall in elderly, and strategies of fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* community dwelling adults without medical conditions to impair walking ability

Exclusion Criteria:

* cognitively or physically unable to cooperate with the examiner to finish the test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of fall | From date of recruitment until the end of the study, assessed up to 42 months (reported once per year)
  Incidence of fall each year

SECONDARY OUTCOMES:
Kinematics test | From date of recruitment until the end of the study, assessed up to 42 months
  During balance tests, assessing kinematics by using inertia sensors.
Kinetics test | From date of recruitment until the end of the study, assessed up to 42 months
  During balance tests, assessing kinetics by using sEMG (high-density surface EMG).
EEG test | From date of recruitment until the end of the study, assessed up to 42 months
  During balance tests, assessing brain mechanisms by using electroencephalogram (EEG).
fNIRS test | From date of recruitment until the end of the study, assessed up to 42 months
  During balance tests, assessing brain mechanisms by using functional near-infrared spectroscopy (fNIRS).
MRI assessments | From date of recruitment until the end of the study, assessed up to 42 months
  Using functional magnetic resonance imaging to assess brain mechanisms during foot movements.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - National Research Center for Rehabilitation Technical Aids, Beijing, Beijing Municipality
  - National Research Center for Rehabilitation Technical Aids, Beijing

IPD SHARING:
Plan to Share IPD: No